CLINICAL TRIAL: NCT00923052
Title: The Natural History of Solid Organ Cancer Stem Cells (SOCSC)
Status: Terminated | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090079; 09-C-0079; NCT00892060 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2015-05-07

CONDITIONS: Hepatic Cancer; Pancreatic Ductal Cancer; Colorectal Cancer; Breast Cancer; Gastric Cancer
Keywords: Cancer Stem Cells; Biomarkers; Surgery; Solid Organ Cancers; Natural History; Cancer; Solid Organ Cancer; Liver Cancer; Colorectal Cancer; Breast Cancer; Gastric Cancer; Pancreatic Ductal Cancer
MeSH Terms: conditions — Liver Neoplasms; Colorectal Neoplasms; Breast Neoplasms; Stomach Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Background:

* Researchers are trying to learn what causes certain types of cancer to spread to other organs in the body (metastasis). Cancer tumors may produce a very small number of specific cells (cancer stem cells) that cause the tumors to grow in other organs throughout the body.
* By examining cancer tumor tissue, normal tissue, blood, bone marrow, and other body fluids, researchers may determine whether these samples contain cancer stem cells. Cancer stem cells may provide information on whether the cancer will come back or spread before other routine x-ray studies or lab tests indicate its presence.

Objectives:

* To acquire a collection of solid organ cancer stem cells for future study.
* To analyze solid organ cancer stem cells from various types of cancer on a genetic level.
* To determine if solid organ cancer stem cells are present in the blood or bone marrow.

Eligibility:

* Patients 16 years of age and older who have solid organ cancer (cancer in the liver, colon, rectum, anus, pancreas, stomach, breast, skin, muscles, fat, connective tissue, uterus, ovary, cervix, vagina, vulva, or inner lining of the abdomen) or a precancerous growth, and who are scheduled to have a biopsy or surgery to remove the cancer as part of their treatment.

Design:

* This is a prospective trial designed to procure solid organ cancer stem cells before either surgery or biopsy.
* All patients registered to this trial will undergo surgery to extirpate their cancer in the NCI
* Prior to surgery or biopsy, 8 tablespoons of blood will be drawn.
* During the surgery or biopsy, a sample of normal tissue will be removed along with the cancerous or precancerous tissue. If separate consent is given, samples of bone marrow will also be taken.
* After discharge, patients will return to the clinic for routine visits every month for the first 3 months following surgery, and then about every 3 months for 2 years, and then every 6 months for 3 years. During the visits, patients will have routine blood and imaging studies done, and researchers will take additional blood samples (about 8 tablespoons at each visit) and optional bone marrow samples (4 teaspoons every 6 months) to be used for research.

DETAILED DESCRIPTION:
Background:

* Traditional models of cancer metastasis posit that cancer metastases might originate stochastically in any cancer cell while, the Cancer-Stem-Cell hypothesis suggests that the metastasizing cells are Solid Organ Cancer Stem Cells (SOCSC).
* SOCSC are relatively resistant to current cancer therapies. Thus, effective treatment for metastatic cancers might require the targeting of SOCSC.
* Knowledge on SOCSC is chiefly derived from cell lines. However, data suggest vast differences between cell lines and SOCSC obtained from fresh tumors.
* This protocol is designed to facilitate fresh tissue procurement to study SOCSC.

Primary Objective:

-To study the natural history of SOCSC from various primary and metastatic solid organ cancers using established phenotypic and functional markers.

Secondary Objectives:

* To analyze SOCSC for potential targets that can be used to design novel cancer therapies that target cancer stem cells.
* To determine whether SOCSC are present in the blood and/or bone marrow, and study their quantitative and/or qualitative changes from time of surgical resection to time of recurrence and/or metastasis.
* To evaluate the potential of SOCSC and their quantitative and/or qualitative changes over time after surgery, to be used in future studies as biomarkers for the early detection of cancer recurrence and/or metastases.
* To collect detailed history, demographic, and treatment data as well as perioperative findings to evaluate potential correlation with the presence or absence of SOCSC.
* To develop an animal model to investigate potential interaction between bone marrow derived stem cells and solid organ cancers.
* To observe the course of normal stem cells over time in patients who had benign tumors that do not show evidence of cancer over time.
* To compare the course of normal stem cells with that of stem cells from patients with solid organ cancers.
* To specifically investigate families with clusters of cancer to determine if there is a relationship between SOCSC and potential familial genetic mutations specific to a particular cancer and if present, to compare these genetic abnormalities with individuals from the same family without cancer.

Eligibility:

* Patients 16 years of age or older with primary or metastatic solid organ cancers requiring resection or other cancer directed therapy that is deemed in the best interest of their cancer care.
* Patients with premalignant neoplasms who are scheduled to undergo surgery or biopsy as part of their diagnostic evaluation.
* Patients must have an ECOG performance score of 0-2.
* Patients must have laboratory and physical examination parameters within acceptable limits by standard of practice guidelines prior to biopsy or surgery.

Design:

* This is a prospective trial designed to procure SOCSC from various benign and solid organ cancers tumors (primary or metastatic) and follow their natural history from time of surgery and or other cancer directed therapy to time of recurrence.
* SOCSC will be isolated using phenotypic and functional markers. Investigations will be performed on the following tissues: Blood prior and after surgery, tumor and adjacent normal tissue when available, bone marrow (strictly optional under separate consent), and peritoneal washings when applicable.
* After surgery blood will be drawn at 1 and 3 months and every 3-6 months thereafter during the follow-up period (5 years). Bone marrow may be analyzed every six months during the follow-up period (strictly optional).
* Patients will be followed with standard of care or other cancer directed therapy deemed in the best interest of the patient.
* It is anticipated that between 274 and 676 patients will be enrolled over a period of 5 years (2-5 patients per month).

ELIGIBILITY:
* INCLUSION CRITERIA: (Beginning with amendment J, all patients must meet the first eligibility criteria a. Patients scheduled to underg

surgery must meet criteria b-e.)

* Patients with radiographic evidence of, biochemical evidence of, and/or histologically/cytologically proven solid organ cancer, including hepatobiliary cancer, pancreatic cancer, colorectal cancer, gastric cancer, breast cancer, adrenal cancer, mesothelioma, anal cancer, female reproductive tract cancer (ovarian, uterine and cervical), melanoma, and sarcoma.
* Patients with rare solid organ cancers including but not limited to small intestine, vagina, vulva, carcinoid, skin, pediatric cancers, Kaposi s sarcoma, and cancers of unknown origin.
* Patients with premalignant neoplasms who are scheduled to undergo surgery or biopsy as part of their diagnostic evaluation.
* Patients with a family history of familial or hereditary solid organ cancers or a clinical suspicion for a familial cancer (these patients may show no evidence of disease at the time of enrollment).
* Patients must have an ECOG performance score of 0-2.
* Patients must be 16 years of age or older.
* Patients must have laboratory and physical examination parameters within acceptable limits by standard of practice guidelines prior to biopsy or surgery. Note: Not applicable for healthy relatives having blood analyzed for DNA only.
* Patients must be seronegative for HIV antibody, Hepatitis B surface antigen and Hepatitis C antibody, with the exception of patients with hepatocellular cancers, who must be seronegative for HIV antibody only. Note: Not applicable for healthy relatives having blood analyzed for DNA only.
* Patients undergoing treatment for their neoplasm under other current NIH protocols may be eligible.

Note: Patients will not undergo surgery or biopsy for the sole purpose of tissue procurement.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2009-02-09; Study Completion 2015-05-07

PRIMARY OUTCOMES:
To study and characterize both quantitatively and qualitatively SOCSC from various primary and metastatic solid organ cancers from time of surgery or other cancer directed therapy to time of recurrence or progression using an exhaustive list of ...

SECONDARY OUTCOMES:
To determine whether SOCSC are present in the blood and/or bone marrow, and study their quantitative and/or qualitative changes over the course of the disease, from time of initial presentation to time of recurrence and/or metastasis.To sp...

CONTACTS AND LOCATIONS:
Overall Officials: Udo Rudloff, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Fidler IJ. Critical factors in the biology of human cancer metastasis: twenty-eighth G.H.A. Clowes memorial award lecture. Cancer Res. 1990 Oct 1;50(19):6130-8. PMID 1698118
- [Background] Fidler IJ. Critical factors in the biology of human cancer metastasis. Am Surg. 1995 Dec;61(12):1065-6. No abstract available. PMID 7486447
- [Background] Fidler IJ. Critical determinants of melanoma metastasis. J Investig Dermatol Symp Proc. 1996 Apr;1(2):203-8. PMID 9627717